CLINICAL TRIAL: NCT01602653
Title: Extracorporeal Shock-wave Therapy for Supraspinatus Calcifying Tendonitis: a Randomized Clinical Trial Comparing Two Different Energy Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Ioppolo, MD, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTJ-2011-0252.R1
Record Dates: First submitted 2012-05-14; First posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Supraspinatus Calcifying Tendonitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): the first group of patients received an energy level of 0.20mJ/mm2, 2400 pulses once a week for 4 weeks.
  Interventions: Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK
- 2 (Active Comparator): The second grouop of patients received 0.10mJ/mm2, 2400 pulses once a week for 4 weeks.
  Interventions: Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK

INTERVENTIONS:
Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK — an energy level of 0.20mJ/mm2, 2400 pulses once a week for 4 weeks.
  Arms: 1
Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK — an energy level of 0.10mJ/mm2, 2400 pulses once a week for 4 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare two different ranges of energy flux density with Extracorporeal Shock Wave Therapy in treatment of supraspinatus calcifying tendonitis.

ELIGIBILITY:
Inclusion Criteria:

* no visible clinical benefits by previous conservative treatment
* medium and large calcific deposits, according to Bosworth classiﬁcation
* type I and II Gartner deposits

Exclusion Criteria:

* presence of tiny calcific deposits, according to Bosworth classiﬁcation
* type III, according to the Gartner classification
* age (if less than 18 years old), diabetes, coagulation diseases or anticoagulant therapy, tumors, bone infections, previous shoulder surgery, pregnancy, pace-maker, acute bursitis demonstrated by ultrasound imaging, rheumatoid arthritis or other connective tissue diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Constant Murley Scale | Change in the mean Constant Murley Scale (CMS) scores at 3 and 6 months was the primary endpoint.
  Constant-Murley scale is the scoring system used to assess shoulder function in four of the studies being reviewed. It combines physical examination tests with subjective evaluations by the patients and consists of 35 points and 65 points respectively. Its strength is the method of its application, which is quite clearly described, and its being an improvement on pre-existing scales

SECONDARY OUTCOMES:
Visual Analogic Scale | The change in the mean Visual Analogic Scale scores from baseline to 3 and 6 months after the intervention
  It is a horizontal line, 10 cm in length with 0 cm labeled "no pain" and 10 cm labeled "worst pain I have ever had". The patient marks on the line the point that they feel represents their perception of their current state

REFERENCES:
- [Derived] Ioppolo F, Tattoli M, Di Sante L, Attanasi C, Venditto T, Servidio M, Cacchio A, Santilli V. Extracorporeal shock-wave therapy for supraspinatus calcifying tendinitis: a randomized clinical trial comparing two different energy levels. Phys Ther. 2012 Nov;92(11):1376-85. doi: 10.2522/ptj.20110252. Epub 2012 Jun 28. PMID 22745199